CLINICAL TRIAL: NCT02814474
Title: Impact of Ketone Bodies on Myocardial Glucose and Fatty Acid Metabolism in Healthy Volunteers: A Positron Emission Tomography Study
Brief Title: Effects of Experimental Hyperketonemia on Myocardial Metabolism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1-10-72-104-14
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
Keywords: PET/CT; Heart failure; hydroxybutyrate
MeSH Terms: conditions — Heart Failure | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SALINE (Placebo Comparator): Infusion of saline (0.9 %)
  Interventions: Other: Saline
- KETONE (Experimental): Infusion of Na-3-Hydroxybutyrate (0.18 g/kg/hour) for 390 minutes
  Interventions: Other: Na-3-hydroxybutyrate

INTERVENTIONS:
Other: Na-3-hydroxybutyrate — Infusion of Na-3-hydroxybutyrate (0.18 g/kg/hour) for 390 minutes
  Arms: KETONE
Other: Saline — Infusion of 0.9 % saline
  Arms: SALINE

SUMMARY:
Starvation and metabolic stress increase circulating ketone bodies, potentially providing the heart with an alternative oxidative fuel. Hyperketonemia reduces myocardial fatty acid consumption. It is unclear whether this is due to inhibited peripheral lipolysis or diminished uptake per se.

Aim: To test whether infusion of 3-hydroxybutyrate (BHB) inhibits myocardial glucose and fatty acid uptake.

Methods: Randomized, single blinded, cross-over interventional study in 8 healthy volunteers. Myocardial glucose and fatty acid metabolism studied by 11C-palmitate and 18F-FDG PET/CT. Experimental elevation of circulating ketone bodies by infusion of β-hydroxy-β-methylbutyrate.

DETAILED DESCRIPTION:
Background:

Ketone bodies are produced by the liver in conditions of increased fatty acid oxidation, serving as important fuel sources during fasting and starvation. They are metabolized to acetyl-CoA which enters the tricarboxylic acid cycle, enabling ATP production independently of glycolysis and resulting in lower oxygen consumption per mole of produced ATP compared to glucose [ref]. Their primary physiological function appears to be as an alternative protein-sparing source of energy for extrahepatic tissues in times of reduced carbohydrate availability, preventing muscle wasting. The principal ketone bodies in humans are beta-hydroxybutyrate (BHB) and acetoacetate. Increased ketogenesis is a feature common to fasting, starvation and diabetes mellitus. Ketones have been shown to have a number of neuroprotective effects including anticonvulsant activity, improving cognitive function in Alzheimer's disease and decreasing the effects of acute brain injury and ischemic damage [ref], as well as antitumoral effect in gliomas. This has led to the suggestion that ketones could be used therapeutically for a number of diseases though currently the only recognized therapeutic use of ketones is in the form of ketogenic diets for the treatment of epilepsy.

There are limited in vivo studies on the effect of ketones on the heart. It is known that fatty acids are the preferred myocardial fuel substrate and that this shifts to increased use of glucose, and to a lesser extent ketones, in times of acutely increased demand. Interestingly, acute ketone infusion in pigs appears to inhibit myocardial fatty acid oxidation. In vitro studies suggest ketones decrease myocardial glucose uptake and affect myocardial contractility, with either increased or decreased contractility when ketones are the only energy source. This has not been further investigated in vivo. It is therefore unclear to what extent ketones can contribute to myocardial metabolism in conditions of hyperketonemia, and how this affects contractility.

The present project thus proposes to address the issues outlined above, by measuring human cerebral and cardiac uptake of energy substrates, together with functional parameters, using PET imaging and appropriate radiotracers, under experimental hyperketonemia.

Hypotheses:

1. An acute increase in blood ketone concentration without previous ketoadaptation will decrease cardiac palmitate and glucose uptake in healthy humans.

Materials and methods

Effect of acute ketone infusion on cardiac perfusion and 18F-FDG and 11C-palmitate uptake in healthy subjects:

Study population: 10 healthy volunteers. All study subjects will be instructed to follow a standardised diet for 1 week before the study. On the study day, they will undergo a baseline dynamic cardiac PET scan with 15O-water followed by 11C-palmitate and 18F-FDG tracers, together with baseline blood samples, muscle biopsy and subcutaneous fat biopsy to assess peripheral metabolic status. An intravenous infusion of sodium betahydroxybutyrate will then be initiated at a concentration and rate sufficient to achieve 1-2 mM ketonemia after 30 minutes (assessed by blood sample). A second dynamic PET scan identical to the first will then be performed under continuous ketone infusion at a constant rate. Finally, a second set of blood samples, muscle and subcutaneous fat biopsies will be taken after the scan before stopping the ketone infusion.

Perspectives:

The results of this research are expected to provide insights into how human heart metabolism respond to increased ketone bodies, and whether there are significant functional improvements. It should contribute to further understanding the possible therapeutic benefits of both exogenous ketone administration and of fasting in relation to cardiac function, with implications for the treatment of various diseases such as diabetes and heart failure. Knowledge of ketones' effects on the kinetics of various radionuclide tracers also has importance for the appropriate clinical use of diagnostic PET scans in patients with elevated blood ketone levels. In addition, the implementation and validation of a ketone PET tracer will allow further future non-invasive studies that directly measure ketone metabolism in various tissues and disease states.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Decreased cardiac function
* Kidney disease
* Pulmonary disease
* Current malignant disease
* Substance abuse
* Blood donation within 6 month prior to the study
* Participation in studies involving ionising radiation within 12 month prior to the study
* Known claustrophobia

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Myocardial Glucose uptake | After 330 minutes of ketone infusion
  Dynamic 18F-FDG PET/CT scan - 50 minutes
Myocardial Fatty Acid Metabolism | After 210 minutes of ketone infusion
  Dynamic 11C-palmitate PET/CT scan - 50 minutes
Myocardial Blood Flow | After 180 minutes of ketone infusion
  Dynamic 15O-H2O PET/CT scan - 6 minutes

SECONDARY OUTCOMES:
Insulin sensitivity | Time 0-390 of the ketone body infusion
  Glucose infusion rate (GIR) during a 0.3 mIE/kg/min hyperinsulinemic- euglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, MD DMsc, Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Nuclear Medicine & PET Center, Aarhus University Hospital, Aarhus
  - Medical Research Laboratories, Aarhus

REFERENCES:
- [Derived] Svart M, Gormsen LC, Espersen R, Rittig N, Starup-Linde J, Moller N, Rejnmark L. 3-Hydroxybutyrate administration elevates plasma parathyroid hormone in a pilot human randomized, controlled, cross over trial. Bone. 2021 Dec;153:116166. doi: 10.1016/j.bone.2021.116166. Epub 2021 Aug 28. PMID 34464780
- [Derived] Lauritsen KM, Sondergaard E, Luong TV, Moller N, Gormsen LC. Acute Hyperketonemia Does Not Affect Glucose or Palmitate Uptake in Abdominal Organs or Skeletal Muscle. J Clin Endocrinol Metab. 2020 Jun 1;105(6):dgaa122. doi: 10.1210/clinem/dgaa122. PMID 32161953
- [Derived] Lauritsen KM, Sondergaard E, Svart M, Moller N, Gormsen LC. Ketone Body Infusion Increases Circulating Erythropoietin and Bone Marrow Glucose Uptake. Diabetes Care. 2018 Dec;41(12):e152-e154. doi: 10.2337/dc18-1421. Epub 2018 Oct 16. No abstract available. PMID 30327354